CLINICAL TRIAL: NCT00627081
Title: Intravenous Opioid-sparing Effect of Thoracic Epidural Administration of Chirocaine (5 mg/ml) During Thoracotomy
Brief Title: Effect of Thoracic Epidural Analgesia on Intravenous Closed-Loop Anesthesia
Acronym: Drone-APDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007/11
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): general anesthesia and thoracic epidural administration of saline
  Interventions: Drug: remifentanil
- 2 (Active Comparator): general anesthesia and thoracic epidural administration of chirocaine
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — dosage
  Other Names: Remifentanil: Ultiva

SUMMARY:
The association of general anesthesia and of thoracic epidural anesthesia is used in thoracic surgery with a demonstrated benefit on the risk of postoperative respiratory complications.

The objective of the study is to analyze the influence of thoracic epidural administration of chirocaine (5 mg/ml) on the administration of anesthetic agents (propofol and remifentanil), these drugs being administrated using a closed-loop system with the Bispectral Index as the controller.

Two groups of patients are compared:

* one group will receive general anesthesia and thoracic epidural administration of saline. Chirocaine will be administered before patient's awakening,
* one group will receive general anesthesia and thoracic epidural administration of chirocaine (5 mg/ml).

In both groups, the closed-loop system ensures that le depth of anesthesia is similar in both groups.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing a thoracotomy under general anesthesia and epidural anesthesia

Exclusion Criteria:

* age lower than 18 years,
* pregnant woman,
* psychotropic treatment,
* central neurological disorder or lesion cerebral,
* allergy to propofol or to a muscle relaxant,
* refusal or contra-indication of epidural anesthesia,
* severe emphysema,
* coronary disease,
* treatment with a beta-blocker or a vasoactive drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
amount of remifentanil delivered by the closed-loop system | end of anesthesia

SECONDARY OUTCOMES:
amount of propofol delivered by the closed-loop system | end of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch, 92150 Suresnes, France
Locations (1):
- Hôpital Foch, Suresnes, France

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963